CLINICAL TRIAL: NCT05629065
Title: Pathways to Advance Targeted and Helpful Serious Illness Conversations (PATH-SIC)
Acronym: (PATH-SIC)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Manz, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 22-501
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Gastrointestinal Cancer; Gynecologic Cancer; Thoracic Cancer; Genitourinary Cancer
Keywords: Breast Cancer; Gastrointestinal Cancer; Gynecologic Cancer; Thoracic Cancer; Genitourinary Cancer; Serious Illness Communication
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms

STUDY DESIGN:
Intervention Model Description: 4 arm randomized clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Both patient and clinician receive a nudge (Experimental): * Patient nudge consists of a letter and SHARE questionnaire
  * Clinician "nudge" email encouraging discussion to initiate discussion on SIC
  Interventions: Other: Clinician Nudge Email; Other: Patient Nudge Letter and Share questionaire
- Neither the patient nor clinician receive a nudge (No Intervention): Standard Care
- Patient receives a nudge but not the clinician (Experimental): -Patient nudge consists of a letter and SHARE questionnaire
  Interventions: Other: Patient Nudge Letter and Share questionaire
- Clinician receives a nudge but not the patient (Experimental): -Clinician "nudge" email encouraging discussion to initiate discussion on SIC
  Interventions: Other: Clinician Nudge Email

INTERVENTIONS:
Other: Clinician Nudge Email — -Clinician "nudge" email encouraging discussion to initiate discussion on SIC at next visit
  Arms: Both patient and clinician receive a nudge; Clinician receives a nudge but not the patient
Other: Patient Nudge Letter and Share questionaire — Involves patient nudge consists of a letter and SHARE questionnaire
  - patient nudge is a letter and a SHARE questionnaire encourages the participant to complete the SHARE questionnaire, which asks questions about the participants goals and preferences around cancer care, and discuss the questionnaire with their oncology clinician at the next visit.
  Arms: Both patient and clinician receive a nudge; Patient receives a nudge but not the clinician

SUMMARY:
The purpose of this study is to increase serious illness conversations (SICs) about patients goals and preferences regarding their healthcare between patients with cancer and their oncology clinicians and improved care provided near the end of life.

DETAILED DESCRIPTION:
The objective of this study is to implement an intervention in a pragmatic randomized controlled trial that uses cancer treatment pathways data to identify patients appropriate for serious illness conversations (SICs) and applies "nudges" to patients and their oncology clinicians to increase SICs and improve end of life (EOL) outcomes.

Identified participants and clinicians will be randomized into 1 or 4 groups.

* Nudge to patient and clinician
* Nudge to patient only
* Nudge to clinician only
* No nudge.

The expected enrollment is approximately 800 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged 18 years or older, reach one of the poor prognosis nodes identified and have an upcoming appointment at one of the following Dana Farber Cancer Institute oncology clinics (including Longwood and Chestnut Hill locations)
* Breast Oncology Clinic
* Gastrointestinal Oncology Clinic
* Genitourinary Oncology Clinic
* Gynecologic Oncology Clinic
* Thoracic Oncology Clinic

Exclusion Criteria:

* Patients with an SIC documented in the Advance Care Planning module of the electronic health record in the 6 months prior to reaching a poor prognosis node
* Patients who have previously been randomized in this trial (e.g., the patient is encountering a poor-prognosis node for the second time during the trial period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an SIC at 60 days for arm 1 (patient +clinician nudge) vs arm 2 (no nudge). | up to 60 days after reaching the poor prognosis node
  The numerator includes patients with any SIC documentation extracted from the Advanced Care Planning module between the date of the poor prognosis node and 60 days. The denominator is all patients randomized to the applicable study arm.

SECONDARY OUTCOMES:
Proportion of patients with an SIC at 60 days, comparison of all 4 study arms | up to 60 days after reaching the poor prognosis node
  Same as the primary outcome
Time from SIC to death among decedents | randomization up to 1 year
  Time from SIC to death among decedents
Receipt of chemotherapy in last 14 days of life | randomization up to 1 year
  Whether or not the patient received chemotherapy in the last 14 days of life, among decedents
ED visits in the last 30 days of life | randomization up to 1 year
  Number of ED visits in the last 30 days of life, among decedents
Hospitalization in last 30 days of life | randomization up to 1 year
  Hospitalization in the last 30 days of life, among decedents
Median length of hospitalization | randomization up to 1 year
  Median length of last hospitalization, in days among decedents
ICU utilization in last 30 days of life | randomization up to 1 year
  ICU hospitalization in the last 30 days of life, among decedents
Death in an acute care facility | randomization up to 1 year
  Presence or absence of death in an acute care facility like a hospital or emergency room
Death in the ICU | randomization up to 1 year
  Whether or not death occurred in an ICU
Hospice enrollment at death | randomization up to 1 year
  Whether or not the patient was enrolled in hospice on the day of death
Enrolled < 4 days in hospice at death | randomization up to 1 year
  Whether or not the patient was enrolled in hospice for less than 4 days on the day of death
Patient preferences | Up to 60 days after randomization
  Patient responses on SHARE questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Manz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu